CLINICAL TRIAL: NCT05695365
Title: Feasibility of Resistance Exercise to Treat Major Depression Via Cerebrovascular Mechanisms: A Pilot Trial
Brief Title: Feasibility of Resistance Exercise to Treat Major Depression Via Cerebrovascular Mechanisms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iowa State University (Other)
Responsible Party: Principal Investigator, Jacob Meyer, Assistant Professor of Kinesiology, Iowa State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-452
Record Dates: First submitted 2022-12-14; First posted 2023-01-25 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Major Depressive Disorder
Keywords: Resistance Exercise
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Resistance Exercise Training (Experimental): Participants will complete a 16-week, twice/week program to increase strength.
  Interventions: Behavioral: Resistance Exercise Training

INTERVENTIONS:
Behavioral: Resistance Exercise Training — Participants will complete a 16-week, twice/week supervised resistance exercise training program to increase strength. Each session will last ~60 minutes and begin and end with a 5-minute aerobic warm-up/cool-down on a cycle ergometer, elliptical, treadmill, or walked laps. Training will begin with a 1-week standard familiarization process to introduce participants to the machines, teach correct lifting techniques, and ensure participant safety and comfort with each exercise machine. Participants will perform 3 sets of 8-12 repetitions on 10 Keiser resistance machines (i.e., leg press, hamstring curl, quadriceps extension, chest press, lat pulldown, shoulder press, biceps curl, triceps extension, abdominal crunch), with a 1-minute rest time between each set. Workload will begin at 50% of the estimated 1-RMs and increase by 5-10% after any session in which a participant completes 12 repetitions in all 3 sets. The workload will be tailored based on progressive increases in strength.

SUMMARY:
This project is a single-arm pilot trial to investigate the feasibility, acceptability, and plausible efficacy of a 16-week resistance exercise training (RET) program for treatment of major depressive disorder.

DETAILED DESCRIPTION:
Resistance exercise training (RET) is a promising but understudied approach for treatment of major depressive disorder (MDD). The purpose of this study is to assess the feasibility of recruiting eligible participants, enrolling them into the study, and retaining them across 16 weeks of resistance exercise training (RET) twice per week for treatment of depression. The primary aim of this study is to determine the feasibility (i.e., recruitment and enrollment rates) and acceptability (i.e., adherence rate, retention rate, and participant satisfaction) of running a larger study that would evaluate the efficacy of RET for treating Major Depressive Disorder (MDD). Secondary aims are to implement and examine the utility of theory-informed adherence strategies (i.e.,exercise preparation habit development and ratings, commitment contracts, and intrinsic motivation reflections) for promoting adherence to exercise sessions, explore efficacy of RET for treating MDD, and explore cerebrovascular function as a potential mechanism of RET's treatment of depression. As such, investigators will recruit 10 individuals with diagnosed MDD (via the Structured Clinical Interview for Depression) and enroll participants in a 16-week RET program. Assessments of depression, cerebrovascular functioning, physical activity, and health will be completed at weeks 0, 8, 16, with a 26-week follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Be diagnosed with DSM-5 (Diagnostic and Statistical Manual of Mental Disorders) MDD confirmed via Structured Clinical Interview for DSM-5
* Have current depressive symptoms of at least mild severity defined by a Hamilton Rating Scale of Depression score greater than or equal to 8
* Be ages 18-65
* Have not changed psychological treatments (including drugs, behavioral and psychological treatments) in the past 8 weeks and willing to maintain treatments throughout study enrollment
* Safe to exercise based on Physical Activity Readiness Questionnaire (PARQ) responses

Exclusion Criteria:

* Currently pregnant, nursing, or planning to become pregnant during the study
* Currently diagnosed with a drug or alcohol use disorder (via SCID)
* Comorbid psychiatric conditions confirmed via SCID, with the exception of Generalized Anxiety Disorder (GAD; due to high comorbidity)
* Class II or greater level of obesity (BMI greater than or equal to 35)
* High active suicidal ideation with specific plan and intent ('4' or '5' score on Suicidal Ideation from Columbia Suicide Severity Rating Scale or '3' on QIDS)
* Currently meets US resistance exercise recommendations per week (2 days per week) for the last 8 weeks
* Self-reported prior cardiovascular event or condition, stroke or pulmonary, renal, or neurological disease
* Self-reported diabetes mellitus
* Self-reported recent (within 3 months) severe concussion, in which the individual lost consciousness for any amount of time
* Self-reported smoking/vaping

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
Recruitment and enrollment rates (feasibility) | Week 26
  Screening responses and timestamps will be used to assess the success of recruitment strategies and recruitment rate, calculated by taking the total number of participants recruited (i.e., completed screening survey) divided by the recruitment period duration. Enrollment rate will be calculated by taking the total number of participants enrolled divided by the recruitment period duration.
Participant satisfaction (acceptability) | Week 26
  Participant satisfaction will be assessed using a mixed-method approach, capturing self-reported ratings of satisfaction with the RET program (six questions regarding satisfaction with responses ranging from 0-46, with higher scores indicating greater level of satisfaction) corroborated by a qualitative semi-structured interview, with responses analyzed using a thematic qualitative analysis.
Retention (acceptability) | Week 26
  The retention rate will be calculated based on the percentage of participants that complete all study visits.
Adherence (acceptability) | Week 26
  The adherence rate will be calculated based on the percent of total study visits (i.e., assessment visits and RET sessions) completed within +/-7 days of the scheduled visit date for each participant.
Change in exercise preparation habit ratings | Change from week 1 habit ratings at week 16
  To facilitate exercise adherence, participants will develop exercise preparation habit action and coping plans during their baseline visit. These plans will subsequently be assessed weekly during exercise sessions, with participants responding to 3 questions regarding their success in developing exercise preparation habits. Using a 5-point Likert scale ranging from "Never" to "Every Time", participants will report 1) how well they were able to stick to their exercise preparation habit action and coping plans, 2) carried through with preparation steps when their identified cue was encountered, and 3) completed the habit without the planned cue. They were also provided an opportunity to revise their habit action and coping plan if their current plan was not successful the previous week.
Change in level of commitment | Change from week 1 level of commitment at week 16
  Participants will be asked to report their current level of commitment to the 16-week program and attending their next exercise session via a visual analogue scale anchored with "0" (0% committed) to "100" (100% committed). They subsequently responded to free-text questions related to what they needed to do or what the research team could do to increase their level of commitment. Next, they answered the question "Will you attend your next RET session?" (yes/no response buttons), and then provided an electronic signature confirming they would attend.
Change in depression symptom severity via GRID-Hamilton Depression Rating Scale (HAM-D) | Change from baseline depression severity at the final assessment
  The GRID-HAM-D is a clinician-completed questionnaire that will be used to rate depressive symptom severity. The questionnaire is designed for adults and is used to rate the intensity and frequency of depressive symptoms by probing mood, feelings of guilt, suicidal ideation, insomnia, agitation or retardation, anxiety, weight loss, and somatic symptoms. Clinical Interviewers will follow the Structured Interview Guide and use GRID scoring, in which dimensions of intensity and frequency of a symptom are rated independently for each item. Higher scores reflect greater symptom severity, categorized as Normal (0-7), Mild Depression (8-13), Moderate Depression (14-18), Severe Depression (19-22), and Very Severe Depression (>23).
Change in depression diagnosis via Structured Clinical Interview for DSM-5 Disorders (SCID) | Change from baseline depression diagnosis at the final assessment
  This is a clinician-administered semi-structured interview guide for making diagnoses according to the diagnostic criteria published in the American Psychiatric Association's Diagnostic and Statistical Manual for Mental Disorders (DSM-5). It provides diagnoses for depressive and bipolar disorders, schizophrenia spectrum and other psychotic disorders, substance use disorders, anxiety disorders (panic disorder, agoraphobia, social anxiety disorder, generalized anxiety disorder), obsessive-compulsive disorder, posttraumatic stress disorder, attention-deficit/hyperactivity disorder, and adjustment disorder. The SCID will be administered by a Clinical Interviewer to diagnose Major Depressive Disorder and assess for exclusion criteria in this study.
Change in depressive symptoms severity via the Quick Inventory of Depressive Symptoms (QIDS) | Change from baseline depression symptoms severity at the final assessment
  This is a self-administered 16-item questionnaire that assesses the severity of nine depressive symptoms in the last 7 days. Each item is rated on a 4-point scale (0-3), with total scores ranging from 0-27. Higher scores indicate more severe depression.
Change in Transcranial Doppler ultrasound of Middle Cerebral Artery (MCA) blood flow velocity | Change in baseline blood flow velocity at the final assessment
  Middle Cerebral Artery (MCA) blood flow velocity will be measured under supine, resting conditions using non-invasive techniques following 10 min of quiet rest in a dimly lit room. It will be assessed in duplicate and averaged for analyses. Measurements will be taken from the left middle cerebral artery (MCA) following standardized, recommended insonation protocols using a 2-MHz Transcranial Doppler (TCD) probe secured to the temporal window via a headset. MCA mean blood velocity will be calculated using a standard algorithm implemented on the device, averaged over a 60-sec epoch.
Change in Transcranial Doppler ultrasound of Middle Cerebral Artery (MCA) blood flow pulsatility | Change in baseline blood flow pulsatility at the final assessment
  Middle Cerebral Artery (MCA) blood flow pulsatility will be measured under supine, resting conditions using non-invasive techniques following 10 min of quiet rest in a dimly lit room. It will be assessed in duplicate and averaged for analyses. Measurements will be taken from the left middle cerebral artery (MCA) following standardized, recommended insonation protocols using a 2-MHz Transcranial Doppler (TCD) probe secured to the temporal window via a headset. Cerebral pulsatility will be quantified using the pulsatility index, calculated as (systolic -diastolic velocity)/mean velocity using TCD, averaged over a 60-sec epoch.

SECONDARY OUTCOMES:
Columbia-Suicide Severity Rating Scale (CSSRS) | Weeks 0, 8, 16, 26
  This is a clinician-administered questionnaire regarding suicidal ideation and behavior. The severity of the ideation subscale is rated on a 5-point ordinal scale: 1 = wish to be dead, 2 = nonspecific active suicidal thoughts, 3 = suicidal thoughts with methods, 4 = suicidal intent, and 5 = suicidal intent with a plan. Suicide behavior is rated on a nominal scale that includes actual, aborted, and interrupted attempts; preparatory behavior; and non-suicidal, self-injurious behavior.
Estimated 1 Repetition Maximum (RM) Strength Test | Weeks 0, 8, 16, 26
  A 5-RM testing method will be used to calculate each participant's estimated 1-RM, in which participants will lift the maximum amount of weight that can be lifted five times with correct form, timing, and breathing. Maximum strength will be assessed on one upper body (chest press) and one lower body (leg press) major muscle group, completed using the Keiser resistance machines.
Grip Strength | Weeks 0, 8, 16, 26
  A research assistant will ask the participant to sit in a chair and rest his/her arm on the table with the elbow on top of a mouse pad and arm held at a right angle to adjust the dynamometer to the participant's hand size. The participant will then squeeze the dynamometer twice to practice. To begin the assessment, the participant will use his/her right hand and squeeze as hard as possible. Three trials will be attempted with each hand. When the right hand is complete, the left hand will be assessed (i.e., 3 trials). A sum of the greatest effort (number) for each hand is totaled (rounded to the nearest 2 kilograms) and will be recorded.
Arterial Stiffness | Weeks 0, 8, 16, 26
  Aortic stiffness will be assessed via carotid-femoral pulse wave velocity (CfPWV). Carotid and femoral pressure waveforms will be captured with applanation tonometry and simultaneous R-wave gating. CfPWV will be calculated as the distance between carotid and femoral sites divided by the time lag (Δt) between carotid-femoral waves.
Carotid Structure | Weeks 0, 8, 16, 26
  The carotid structure will be assessed by measuring diameter, wall thickness, and stiffness using ultrasound and carotid pressures obtained from contralateral carotid tonometry during CfPWV assessment. WV-β will be calculated using onboard wall-tracking software to determine common carotid stiffness and diameter. Carotid wall thickness (IMT) will be measured using semi-automated calipers.
International Physical Activity Questionnaire Short Form | Weeks 0, 8, 16, 26
  The International Physical Activity Questionnaire Short Form (IPAQ-SF) is a measure that assesses the types of the intensity of physical activity and sitting time that people did over the past 7 days using seven questions via self-report by the participant. Participants are instructed to report the number of days per week and minutes per day they spend engaging in 1) vigorous activity, 2) moderate activity, 3) walking, and 4) sitting. Responses are used to calculate total minutes of walking, minutes of moderate-to-vigorous physical activity per week, and hours of sitting time on a weekday and weekend day, with higher scores indicating greater levels of each behavior.
activPAL (sedentary time and MVPA) | Monitors worn for 7 days following week 0 (intake assessment) and 7 days prior to week 8 and 16 assessments
  Participants will place an activPAL on the midline of the thigh on either leg and wear the monitor 24 hours per day, removing it only for water-based activities (e.g., swimming). For data to be valid, the monitor must have been worn for 20 hours on at least 4 days, including a minimum of 3 weekdays and 1 weekend day. Sleep time will be parsed out from each day's sitting/lying time automatically using PALanalysis. From these data, average minutes of sitting per day will be used to assess total sedentary time, minutes of stepping time with a cadence ≥75 and <100 will be used to assess minutes of light intensity physical activity, and minutes of stepping time with a cadence ≥100 will be used to assess minutes of moderate to vigorous physical activity (MVPA).
36-Item Short Form Health Survey (SF-36) | Weeks 0, 8, 16, 26
  The SF-36 assesses health-related qualify of life. It consists of eight scaled scores (including vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning, and mental health), which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability (i.e., a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability).
Penn State Worry Questionnaire (PSWQ) | Weeks 0, 8, 16, 26
  The Penn State Worry Questionnaire (PSWQ) is a 16-item questionnaire that assesses the trait of worry, using Likert rating from 1 (not at all typical of me) to 5 (very typical of me). The total scores range from 16 to 80 with higher scores indicating greater levels of worry.
Perceived Stress Scale (PSS-10) | Weeks 0, 8, 16, 26
  This is a 10-item questionnaire to measure an individual's level of perceived stress in the past month. The response options for each feeling or thought indicate the frequency with which it occurred: 0 = Never; 1 = Almost Never; 2 = Sometimes; 3 = Fairly Often; 4 = Very Often.
Exercise Identity Scale (EIS) | Weeks 0, 8, 16, 26
  The EIS is a 9-item questionnaire used to assess the salience of identifying with exercise as an integral portion of the self-concept. Participants respond to each EIS item on a scale, anchored by (1) Strongly Disagree and (7) Strongly Agree, after reading a stem that contextualized each item within their personal exercise experiences (e.g., "The following questions concern your personal beliefs about exercise. Please indicate the degree to which you agree or disagree with each statement when thinking about your exercise participation."). Higher scores reflect greater feelings of exercise as an integral part of their self-identity.

CONTACTS AND LOCATIONS:
Locations (1):
- Iowa State University, Ames, Iowa, United States

IPD SHARING:
Plan to Share IPD: No
There are no known plans for future use.

REFERENCES:
- [Derived] Meyer JD, Perkins SL, Gidley JM, Kuzniar JM, Phillips LA, Lansing JL, Wade NG, Herring MP, Lefferts WK. Feasibility and preliminary efficacy of a theory-informed resistance exercise training single-arm intervention for major depression. Psychol Sport Exerc. 2024 Jul;73:102642. doi: 10.1016/j.psychsport.2024.102642. Epub 2024 Apr 12. PMID 38615899